CLINICAL TRIAL: NCT00225186
Title: A Multi-center, Open, One-arm Study to Investigate the Safety and Efficacy of Daily Oral Administration of T00660AA for the Treatment of Endometriosis Over 52 Weeks (Follow-up to Study 307041)
Brief Title: Safety and Efficacy of SH T00660AA in Treatment of Endometriosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91234; 307059 (Other: company internal)
Record Dates: First submitted 2005-09-22; First posted 2005-09-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Visanne (SH T00660AA , BAY86-5258)

INTERVENTIONS:
Drug: Visanne (SH T00660AA , BAY86-5258) — Daily long-term drug treatment (12 months), and post-treatment observation (6 months) in a subgroup of patients

SUMMARY:
The purpose of this study is to demonstrate safety and efficacy of SH T00660AA for the treatment of endometriosis

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with endometriosis-associated pelvic pain

Exclusion Criteria:

* Pregnant or lactating women
* History or suspicion of hormone dependent tumor
* Therapy resistant endometriosis or need for primary surgical treatment
* Any other conditions which forbid the participation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2004-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety assessment of the drug | 12-18 months

SECONDARY OUTCOMES:
Efficacy (reduction of pelvic pain) | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (25):
- Germany (17):
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Krumbach, Bavaria
  - München, Bavaria
  - Nuremberg, Bavaria
  - Giessen, Hesse
  - Mühlheim am Main, Hesse
  - Aachen, North Rhine-Westphalia
  - Gevelsberg, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Dippoldiswalde, Saxony
  - Leipzig, Saxony
  - Marienberg, Saxony
  - Weißig, Saxony
  - Kalbe, Saxony-Anhalt
  - Lübeck, Schleswig-Holstein
  - Greifswald
- Italy (5):
  - Brescia
  - Cagliari
  - Napoli
  - Roma
  - Torino
- Ukraine (3):
  - Chernivtsi
  - Kiev
  - Vinnitsa

REFERENCES:
- [Result] Strowitzki T, Faustmann T, Gerlinger C, Seitz C. Dienogest in the treatment of endometriosis-associated pelvic pain: a 12-week, randomized, double-blind, placebo-controlled study. Eur J Obstet Gynecol Reprod Biol. 2010 Aug;151(2):193-8. doi: 10.1016/j.ejogrb.2010.04.002. Epub 2010 May 5. PMID 20444534
- [Result] Kohler G, Faustmann TA, Gerlinger C, Seitz C, Mueck AO. A dose-ranging study to determine the efficacy and safety of 1, 2, and 4mg of dienogest daily for endometriosis. Int J Gynaecol Obstet. 2010 Jan;108(1):21-5. doi: 10.1016/j.ijgo.2009.08.020. PMID 19819448
- [Result] Gerlinger C, Schumacher U, Faustmann T, Colligs A, Schmitz H, Seitz C. Defining a minimal clinically important difference for endometriosis-associated pelvic pain measured on a visual analog scale: analyses of two placebo-controlled, randomized trials. Health Qual Life Outcomes. 2010 Nov 24;8:138. doi: 10.1186/1477-7525-8-138. PMID 21106059
- [Result] Petraglia F, Hornung D, Seitz C, Faustmann T, Gerlinger C, Luisi S, Lazzeri L, Strowitzki T. Reduced pelvic pain in women with endometriosis: efficacy of long-term dienogest treatment. Arch Gynecol Obstet. 2012 Jan;285(1):167-73. doi: 10.1007/s00404-011-1941-7. Epub 2011 Jun 17. PMID 21681516